CLINICAL TRIAL: NCT02231580
Title: A Dose Escalation, Proof of Concept, Phase IIa Study to Investigate the Safety and Tolerability, the Pharmacokinetic and the Pharmacodynamic of BN82451B, Administered Twice Daily Over 4 Weeks, in Male Patients With Huntington's Disease
Brief Title: Study Exploring Safety, Pharmacokinetic and Pharmacodynamic of BN82451 in Male Huntington's Disease Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to subject recruitment problems.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8-55-52966-005; 2013-002899-41 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Huntington's Disease
Keywords: Neurodegenerative genetic disorder
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BN82451B (Experimental): BN82451B capsule: Up to 3 dose levels (40, 60 or 80 mg) twice daily administered orally.
  Interventions: Drug: BN82451B
- Placebo (Placebo Comparator): Placebo capsule: Up to 3 dose levels (40, 60 or 80 mg) twice daily administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BN82451B — BN82451B capsule
  Arms: BN82451B
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of BN82451B versus placebo after oral administration twice daily (bid) for 28 days in patients with Huntington's Disease (HD).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 20 to 70 years old (inclusive).
* Provision of written informed consent prior to any study related procedures. In this study consent may be provided by the legal guardian or carer.
* Confirmed symptomatic Huntington's Disease diagnosed based on clinical features (i.e. Diagnostic Confidence Level equal to 4) and presence of at least 36 cytosine adenine guanine (CAG) repeats in the Huntington gene as documented by a copy of a previous genetic test report.
* Unified Huntington's Disease Rated Scale-Total Motor Score (UDHRS-TMS) greater than or equal to 15.
* Ambulatory.
* UDHRS-Total Functional Capacity (TFC) greater than or equal to 3 (i.e. Shoulson & Fahn Scale stages 1-3 inclusive.
* Subjects on antipsychotic, antidepressant, anxiolytic and hypnotic therapy must have been on stable treatment 4 weeks prior to study drug start and during the study period.
* Able to swallow study medication.
* Able to perform Q-Motor tests.
* If his partner is at risk of pregnancy, the subject agrees to use a condom or be abstinent for 14 days after the last intake of study drug.

Exclusion Criteria:

* Juvenile forms of Huntington's Disease.
* Any form of chorea other than Huntington's Disease.
* History of seizure, epilepsy or other convulsive disorder, with the exception of febrile seizures in childhood.
* History of conditions susceptible to induce seizures such as severe traumatic brain injury, brain tumours, stroke.
* History of neurosurgical procedure.
* Current evidence or history (within 1 year of Baseline) of psychosis, hallucinations or delusions, including major depression with psychotic features, as defined in the Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR). Patients currently experiencing mild depression, or moderate depression which is adequately and appropriately treated in the judgement of the investigator, can participate if depression is not expected to interfere with study participation.
* History of drug and/or alcohol abuse as per the DSM IV-TR criteria within 12 months prior to Baseline.
* At imminent risk of self harm based on investigator's clinical judgment, with a "yes" answer on item 4 or 5 on the Columbia-Suicide Severity Rating Scale (CSSRS) questionnaire.
* Mini Mental State Exam (MMSE) total score less than or equal to 23.
* Used any investigational drugs within 30 days prior to Screening or 5 half lives, whichever is the longest.
* Known allergy/sensitivity to the study drugs or their excipients.
* A severe or ongoing unstable medical condition (e.g. cardiac, hepatic, renal, metabolic or endocrine).
* Any clinically significant condition which, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
* Any significant laboratory results which, in the investigator's opinion, would not be compatible with study participation or represent a risk for subjects while in the study.
* History of malignant disease within the 5 years prior to Screening (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised, in situ prostate cancer with a normal prostate specific antigen).
* An estimated Creatinine Clearance (CrCl) of less than 60 mL/minute (using the Cockcroft-Gault formula).
* Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) values greater than or equal to 2 times the Upper Limit of Normal range (ULN) or both GGT and ALT values greater than three times the ULN.
* Known history of hepatitis B or C or Human Immunodeficiency Virus (HIV) or positive serology at Screening.
* Corrected QT interval using Bazett's correction (QTcB) greater than 450 ms or other clinically significant ECG findings.
* Receiving tetrabenazine within 4 weeks prior to Baseline.
* Taking the following prohibited medications/substances: Strong Cytochrome (CYP) 3A4 inhibitors and Strong CYP3A4 inducers (Wash out prior to Baseline 30 days or 5 half lives,whichever is the longest), CYP2B6 substrates, CYP1A2 substrates, CYP3A4 substrates, CYP2C19 substrates (assessed on a case by case basis)

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Mönchengladbach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a double blind, placebo controlled, randomised, sequential dose ranging repeated dose trial where patients were recruited to a single study centre in Germany. It was planned to enrol 30 patients (10 in each of 3 cohorts). Patients were enrolled to the study from 1 September 2014 until early termination of the study on 31 March 2016.
Pre-assignment Details: Male patients 20-70 years with a documented diagnosis of Huntington's Disease (HD) with at least 36 cytosine adenine guanine repeats in the Huntington gene were screened. Eligibile patients needed to meet defined criteria during quantitative motor function assessments. 25 patients were screened, 17 were enrolled and randomised to treatment.
Groups:
- BN82451B: Patients were randomised to receive oral study medication, BN82451B, b.i.d. from Day 1 to Day 27, under double-blinded conditions. On Day 28 only one morning dose of BN82451B was administered. It was planned for patients to be assigned to 3 cohorts to receive 3 dose levels ranging between 40 and 80 milligrams (mg) b.i.d.
  For cohort 1, 40 mg BN82451B b.i.d. was administered during the first 14 days. If this dose was well tolerated then it was increased to 60 mg b.i.d. for 13 days and one morning dose of 60 mg on Day 28.
  For cohort 2, 60 mg BN82451B b.i.d. was administered during the first 14 days. If 60 mg b.i.d was well tolerated then it was increased to 80 mg b.i.d. for 13 days and one morning dose of 80 mg on Day 28.
  For cohort 3 it was planned to administer 80 mg BN82451B b.i.d for 27 days with one morning dose of 80 mg on Day 28. The study was terminated early before completion of cohort 2.
- Placebo: Patients were randomised to receive oral placebo b.i.d. from Day 1 to Day 27, under double-blinded conditions. On Day 28 only one morning dose of placebo was administered. It was planned for patients to be assigned to 3 cohorts to receive 3 dose levels ranging between 40 and 80 mg b.i.d.
  For cohort 1, 40 mg placebo b.i.d. was administered during the first 14 days. If this dose was well tolerated then it was increased to 60 mg b.i.d. for 13 days and one morning dose of 60 mg on Day 28.
  For cohort 2, 60 mg placebo b.i.d. was administered during the first 14 days. If 60 mg b.i.d was well tolerated then it was increased to 80 mg b.i.d. for 13 days and one morning dose of 80 mg on Day 28.
  For cohort 3 it was planned to administer 80 mg placebo b.i.d for 27 days with one morning dose of 80 mg on Day 28. The study was terminated early before completion of cohort 2.
Period: Overall Study
Arm/Group | BN82451B | Placebo
Started | 14 | 3
Cohort 1 | 8 | 2
Cohort 2 | 6 | 1
Completed | 9 | 3
Not Completed | 5 | 0
Not completed — Adverse Event | 5 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the Safety Population, consisting of all randomised patients who received at least one dose of study medication.
Arm/Group | BN82451B | Placebo | Total Title
Number analyzed (Participants) | 14 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (14.4) | 50.0 (8.7) | 46.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Patients Experiencing Treatment Emergent Adverse Events (TEAEs).
Description: The safety and tolerability of BN82451B versus placebo was determined after oral administration b.i.d. for 28 days in patients with HD. Numbers of patients experiencing TEAEs, including information on seriousness, intensity, drug relationship and those leading to withdrawal are presented for all doses of BN82451B and placebo.
Time Frame: From Day 1 to end of study (a period of up to 7 weeks).
Population: The Safety Population consisted of all randomised patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 14 | 3
Participants
  Patients with any TEAEs | 11 | 2
  Patients with any serious TEAE | 0 | 0
  Patients with at least 1 severe TEAE | 0 | 0
  Patients with at least 1 moderate TEAE | 8 | 1
  Patients with at least 1 mild TEAE | 11 | 1
  Patients with TEAEs related to study medication | 9 | 0
  Patients with TEAEs leading to withdrawal | 5 | 0
  Patients with any TEAEs leading to death | 0 | 0

2. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC)
Description: The AUC was determined for BN82451B and its metabolites BN2468 and BN7167 within a dosage interval (0-12 hours) on Days 1, and 14 and 28. Day 1 data represent the AUC after the first dose (AUC[0-12]). The data for Days 14 and 28 (AUC[τ,ss]) represent the AUC at steady state at the initial cohort dose and following dose escalation, respectively. Data is presented for cohorts 1 and 2, as the study terminated prior to dosing of cohort 3.
Time Frame: 0-12 hours on Days 1, 14 and 28
Population: The PK population consisted of all subjects from the safety population who had no major protocol deviations affecting the PK variables and who had a sufficient number of plasma BN82451B concentrations to estimate the main PK parameters.
Measure: Mean (Standard Deviation); unit: hours*nanograms per millilitre (h*ng/mL)
Groups:
- BN82451B Cohort 1: Patients randomised to receive BN82451B in cohort 1 received doses ranging from 40 to 60 mg BN82451B orally b.i.d. for up to 28 days.
- BN82451B Cohort 2: Patients randomised to receive BN82451B in cohort 2 received doses ranging from 60 to 80 mg BN82451B orally b.i.d. for up to 28 days.
Arm/Group | BN82451B Cohort 1 | BN82451B Cohort 2
Number analyzed (Participants) | 8 | 6
hours*nanograms per millilitre (h*ng/mL)
  Day 1 BN82451B AUC(0-12) | 512.93 (112.53) | 783.78 (144.45)
  Day 1 BN2468 AUC(0-12): number analyzed (Participants) | 8 | 0
  Day 1 BN2468 AUC(0-12) | 90.66 (40.68) |
  Day 1 BN7167 AUC(0-12) | 16.82 (9.01) | 31.67 (24.63)
  Day 14 BN82451B AUCτ,ss | 1521.11 (593.22) | 2594.05 (1077.08)
  Day 14 BN2468 AUC(τ,ss) | 735.51 (203.91) | 1531.00 (412.43)
  Day 14 BN7167 AUC(τ,ss) | 33.39 (20.08) | 46.73 (36.76)
  Day 28 BN82451B AUC(τ,ss) | 2357.95 (977.74) | 3313.45 (1517.6)
  Day 28 BN2468 AUC(τ,ss) | 1509.67 (105.94) | 1936.35 (569.97)
  Day 28 BN7167 AUC(τ,ss) | 34.64 (16.05) | 63.81 (57.70)

3. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Cmax was determined for BN82451B and its metabolites BN2468 and BN7167 on Days 1, 14 and 28. Day 1 data represent the PK after the first dose (Cmax). The data for Days 14 and 28 represent the Cmax at steady state (Cmax,ss) at the initial cohort dose and following dose escalation, respectively. Data is presented for cohorts 1 and 2, as the study terminated prior to dosing of cohort 3.
Time Frame: Days 1, 14 and 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BN82451B Cohort 1 | BN82451B Cohort 2
Number analyzed (Participants) | 8 | 6
ng/mL
  Day 1 BN82451B Cmax | 71.61 (14.81) | 101.45 (16.25)
  Day 1 BN2468 Cmax | 9.03 (4.14) | 18.87 (13.00)
  Day 1 BN7167 Cmax | 3.62 (1.62) | 5.61 (3.62)
  Day 14 BN82451B Cmax,ss | 162.88 (56.31) | 271.64 (99.90)
  Day 14 BN2468 Cmax,ss | 75.34 (15.16) | 125.34 (38.13)
  Day 14 BN7167 Cmax,ss | 4.90 (2.35) | 6.28 (3.55)
  Day 28 BN82451B Cmax,ss | 251.77 (105.64) | 340.41 (156.61)
  Day 28 BN2468 Cmax,ss | 135.19 (5.06) | 171.64 (47.64)
  Day 28 BN 7167 Cmax,ss | 5.51 (1.82) | 9.54 (6.92)

4. Secondary Outcome: Time to Peak Plasma Concentration (Tmax)
Description: Tmax is the empirical time of Cmax and was determined for BN82451B and its metabolites BN2468 and BN7167 on Days 1, 14 and 28. Day 1 data represent the PK after the first dose (Tmax). The data for Days 14 and 28 represent the Tmax at steady state (Tmax,ss) at the initial cohort dose and following dose escalation, respectively. Data is presented for cohorts 1 and 2, as the study terminated prior to dosing of cohort 3.
Time Frame: Days 1, 14 and 28
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BN82451B Cohort 1 | BN82451B Cohort 2
Number analyzed (Participants) | 8 | 6
hours
  Day 1 BN82451B Tmax | 3.0 [2.0 to 3.0] | 2.51 [2.0 to 3.0]
  Day 1 BN2468 Tmax | 9.98 [1.0 to 12.02] | 11.92 [11.92 to 11.92]
  Day 1 BN7167 Tmax | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00]
  Day 14 BN82451B Tmax,ss | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.5]
  Day 14 BN2468 Tmax,ss | 4 [1.05 to 8] | 2.51 [1 to 8]
  Day 14 BN7167 Tmax,ss | 1 [1 to 2.13] | 1 [1 to 2]
  Day 28 BN82451B Tmax,ss | 3 [2.02 to 4] | 2.56 [2 to 3.02]
  Day 28 BN2468 Tmax,ss | 4.06 [2 to 6] | 2.06 [1 to 12]
  Day 28 BN7167 Tmax,ss | 1 [0.55 to 2] | 1.52 [1 to 2]

5. Secondary Outcome: Change From Baseline to Day 28 in the Position-index as Determined by Choreomotography
Description: Choreatic (involuntary) movements were assessed using Choreomotography by calculating a position-index and orientation-index. Patients were asked to grasp and lift a device equipped with an electromagnetic sensor, and were asked to hold the device as stable as possible. Three dimensional (3D) changes in position (x, y and z) and orientation (roll, pitch and yaw) were recorded and used to calculate a position-index and an orientation-index. This method provided an objective measure of the involuntary movements. 5 trials of 20 seconds duration were performed with each hand, and the start and end of each trial was signalled by a cueing tone. The mean changes from Baseline to Day 28 in the position-index of the right and left hands are presented as raw data. The statistical analyses present geometric least squares (GLS) mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: The Pharmacodynamic (PD) population consisted of all subjects from the safety population who have not reported major protocol violations impacting quantitative measures of motor function (Q-motor) evaluation and who have a Q-motor evaluation assessed both at Baseline (Day -1) and at one post baseline visit.
Measure: Mean (Standard Deviation); unit: metres per second (m/s)
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
metres per second (m/s)
  Left hand position-index | 0.021 (0.024) | 0.009 (0.007)
  Right hand position-index | 0.018 (0.014) | 0.009 (0.006)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand position-index statistical analysis is presented (BN82451B versus Placebo). The Mixed Effect Model Repeat Measurement (MMRM) analysis was performed on log-transformed data using the restricted maximum likelihood (REML) model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5743, MMRM; GLS mean ratio = 1.104, 90% CI 2-sided [0.823 to 1.482]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand position-index statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.4349, MMRM; GLS mean ratio = 1.141, 90% CI 2-sided [0.862 to 1.510]

6. Secondary Outcome: Change From Baseline to Day 28 in the Orientation-index as Determined by Choreomotography
Description: Choreatic (involuntary) movements were assessed using Choreomotography by calculating a position-index and orientation-index. Patients were asked to grasp and lift a device equipped with an electromagnetic sensor, and were asked to hold the device as stable as possible. 3D changes in position (x, y and z) and orientation (roll, pitch and yaw) were recorded and used to calculate a position-index and an orientation-index. This method provided an objective measure of the involuntary movements. 5 trials of 20 seconds duration were performed with each hand, and the start and end of each trial was signalled by a cueing tone. The mean changes from Baseline to Day 28 in the orientation-index of the right and left hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: The PD population consisted of all subjects from the safety population who have not reported major protocol violations impacting Q-motor evaluation and who have a Q-motor evaluation assessed both at Baseline (Day -1) and at one post baseline visit.
Measure: Mean (Standard Deviation); unit: radians per second (radians/s)
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
radians per second (radians/s)
  Left hand orientation-index | 0.131 (0.125) | 0.082 (0.100)
  Right hand orientation-index | 0.098 (0.087) | 0.054 (0.045)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand orientation-index statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.8937, MMRM; GLS mean ratio = 1.035, 90% CI 2-sided [0.675 to 1.587]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand orientation-index statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6360, MMRM; GLS mean ratio = 1.093, 90% CI 2-sided [0.800 to 1.493]

7. Secondary Outcome: Change From Baseline to Day 28 in the Mean Grip Force Variability as Determined by Manumotography
Description: The coordination of isometric grip forces in the precision grip between the thumb and index finger were assessed by Manumotography. Grip forces were assessed during grip initiation, object transport and in a static holding phase. Subjects were instructed to grasp and lift a device equipped with a force transducer and 3D position sensor in the precision grip between thumb and index finger and hold it stable adjacent to a marker 10 centimetres high. Grip forces and 3D position and orientation of the object were recorded. Mean isometric grip forces and grip force variability in the static phase (expressed as coefficient of variation = standard deviation/mean x 100 [GFV-C]) were calculated during a 15 second period. 5 trials of 20 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the grip force variability of each hand are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
percentage of variation
  Left hand grip force variability | 5.74 (4.38) | 2.61 (4.57)
  Right hand grip force variability | 5.82 (7.94) | 2.35 (1.17)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand grip force variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2865, MMRM; GLS mean ratio = 1.247, 90% CI 2-sided [0.886 to 1.756]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand grip force variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5338, MMRM; GLS mean ratio = 1.160, 90% CI 2-sided [0.781 to 1.724]

8. Secondary Outcome: Change From Baseline to Day 28 in the Mean Isometric Grip Forces as Determined by Manumotography
Description: The coordination of isometric grip forces in the precision grip between the thumb and index finger were assessed by Manumotography. Grip forces were assessed during grip initiation, object transport and in a static holding phase. Subjects were instructed to grasp and lift a device equipped with a force transducer and 3D position sensor in the precision grip between thumb and index finger and hold it stable adjacent to a marker 10 centimetres high. Grip forces and 3D position and orientation of the object were recorded. Mean isometric grip forces and grip force variability in the static phase (expressed as coefficient of variation = standard deviation/mean x 100 [GFV-C]) were calculated during a 15 second period. 5 trials of 20 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the mean isometric grip forces of each hand are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
Newton
  Left hand isometric grip forces | -0.75 (2.86) | 1.55 (1.99)
  Right hand isometric grip forces | -2.06 (6.00) | 0.91 (1.67)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand isometric grip forces statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0864, MMRM; GLS mean ratio = 0.693, 90% CI 2-sided [0.487 to 0.985]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand isometric grip forces statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0399, MMRM; GLS mean ratio = 0.686, 90% CI 2-sided [0.508 to 0.925]

9. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of Inter Onset Intervals (IOI) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of tap IOI in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of IOI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left finger IOI variability | 0.039 (0.048) | -0.009 (0.002)
  Right finger IOI variability | 0.057 (0.062) | 0.038 (0.049)
  Left finger IOI duration | 0.088 (0.075) | -0.015 (0.041)
  Right finger IOI duration | 0.069 (0.059) | 0.032 (0.031)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0574, MMRM; GLS mean ratio = 1.509, 90% CI 2-sided [1.060 to 2.150]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.8277, MMRM; GLS mean ratio = 0.953, 90% CI 2-sided [0.662 to 1.372]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left finger IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0162, MMRM; GLS mean ratio = 1.238, 90% CI 2-sided [1.074 to 1.426]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right finger IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6320, MMRM; GLS mean ratio = 1.038, 90% CI 2-sided [0.912 to 1.182]

10. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of Tap Durations (TD) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of TD in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of TD for the left and right hands are presented a raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left finger Variability of TD | 0.007 (0.024) | -0.007 (0.015)
  Right finger Variability of TD | 0.017 (0.016) | 0.012 (0.017)
  Left finger Duration of TD | 0.010 (0.021) | -0.011 (0.039)
  Right finger Duration of TD | 0.012 (0.021) | 0.001 (0.025)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger variability of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3005, MMRM; GLS mean ratio = 1.308, 90% CI 2-sided [0.85 to 2.014]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger variability of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.4793, MMRM; GLS mean ratio = 1.177, 90% CI 2-sided [0.804 to 1.722]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left finger duration of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2653, MMRM; GLS mean ratio = 1.150, 90% CI 2-sided [0.934 to 1.416]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right finger duration of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6777, MMRM; GLS mean ratio = 1.045, 90% CI 2-sided [0.875 to 1.248]

11. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of Inter Peak Intervals (IPI) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of tap IPI in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of IPI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left finger IPI variability | 0.040 (0.049) | -0.009 (0.007)
  Right finger IPI variability | 0.057 (0.067) | 0.038 (0.044)
  Left finger IPI duration | 0.088 (0.076) | -0.017 (0.042)
  Right finger IPI duration | 0.069 (0.059) | 0.031 (0.030)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0326, MMRM; GLS mean ratio = 1.618, 90% CI 2-sided [1.124 to 2.331]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6016, MMRM; GLS mean ratio = 0.886, 90% CI 2-sided [0.605 to 1.299]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left finger IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0152, MMRM; GLS mean ratio = 1.242, 90% CI 2-sided [1.077 to 1.433]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right finger IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6033, MMRM; GLS mean ratio = 1.042, 90% CI 2-sided [0.915 to 1.186]

12. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of Inter Tap Intervals (ITI) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of ITI in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of ITI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left finger ITI Variability | 0.041 (0.05) | -0.007 (0.01)
  Right finger ITI Variability | 0.053 (0.068) | 0.03 (0.034)
  Left finger ITI Duration | 0.078 (0.076) | -0.005 (0.006)
  Right finger ITI Duration | 0.056 (0.048) | 0.03 (0.046)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0520, MMRM; GLS mean ratio = 1.657, 90% CI 2-sided [1.086 to 2.529]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6978, MMRM; GLS mean ratio = 0.916, 90% CI 2-sided [0.630 to 1.333]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left finger ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0522, MMRM; GLS mean ratio = 1.298, 90% CI 2-sided [1.043 to 1.614]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right finger ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.9012, MMRM; GLS mean ratio = 1.014, 90% CI 2-sided [0.837 to 1.229]

13. Secondary Outcome: Change From Baseline to Day 28 in the Mean Variability of Peak Tapping Forces (TF) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of TD in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the variability of TF for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
percentage of variation
  Left finger TF | 0.65 (6.97) | -6.43 (6.26)
  Right finger TF | 3.75 (12.86) | -0.11 (8.26)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger TF statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1779, MMRM; GLS mean ratio = 1.198, 90% CI 2-sided [0.96 to 1.494]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger TF statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.8036, MMRM; GLS mean ratio = 0.966, 90% CI 2-sided [0.765 to 1.220]

14. Secondary Outcome: Change From Baseline to Day 28 in the Mean Tapping Frequency (Freq) as Assessed by Digitomotography
Description: Digitomotography was used to assess the duration and the variability of TD in an index finger speeded tapping task. The patient placed their hand on a hand rest with their index finger positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to finger tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The tapping frequency was calculated as the number of taps between the onsets of the first and the last tap divided by the time in between. The mean changes from Baseline to Day 28 in the tapping frequency for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
Hertz
  Left finger freq | -0.492 (0.382) | -0.001 (0.315)
  Right finger freq | -0.466 (0.389) | -0.365 (0.231)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left finger freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0177, MMRM; GLS mean ratio = 0.812, 90% CI 2-sided [0.706 to 0.935]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right finger freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6491, MMRM; GLS mean ratio = 0.967, 90% CI 2-sided [0.856 to 1.093]

15. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of IOI as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of IOI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left hand IOI variability | 0.032 (0.135) | 0.036 (0.023)
  Right hand IOI variability | 0.031 (0.094) | 0.163 (0.276)
  Left hand IOI duration | 0.054 (0.114) | 0.028 (0.043)
  Right hand IOI duration | 0.074 (0.101) | 0.074 (0.132)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6176, MMRM; GLS mean ratio = 1.168, 90% CI 2-sided [0.697 to 1.955]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.4541, MMRM; GLS mean ratio = 0.759, 90% CI 2-sided [0.411 to 1.399]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left hand IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2018, MMRM; GLS mean ratio = 1.119, 90% CI 2-sided [0.967 to 1.294]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right hand IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6527, MMRM; GLS mean ratio = 1.046, 90% CI 2-sided [0.886 to 1.234]

16. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of TD as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of TD for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left hand variability of TD | 0.001 (0.138) | 0.023 (0.026)
  Right hand variability of TD | -0.012 (0.073) | 0.078 (0.128)
  Left hand duration of TD | -0.006 (0.088) | 0.017 (0.027)
  Right hand duration of TD | -0.019 (0.089) | 0.022 (0.069)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand variability of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.8279, MMRM; GLS mean ratio = 0.929, 90% CI 2-sided [0.529 to 1.630]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand variability of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2738, MMRM; GLS mean ratio = 0.612, 90% CI 2-sided [0.292 to 1.283]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left hand duration of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.9218, MMRM; GLS mean ratio = 1.018, 90% CI 2-sided [0.752 to 1.378]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right hand duration of TD statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5032, MMRM; GLS mean ratio = 0.847, 90% CI 2-sided [0.561 to 1.277]

17. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of IPI as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of IPI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left hand IPI variability | 0.045 (0.124) | 0.049 (0.046)
  Right hand IPI variability | 0.027 (0.07) | 0.131 (0.219)
  Left hand IPI duration | 0.057 (0.109) | 0.029 (0.04)
  Right hand IPI duration | 0.079 (0.105) | 0.066 (0.118)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6759, MMRM; GLS mean ratio = 1.140, 90% CI 2-sided [0.677 to 1.917]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5764, MMRM; GLS mean ratio = 0.815, 90% CI 2-sided [0.444 to 1.496]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left hand IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2127, MMRM; GLS mean ratio = 1.115, 90% CI 2-sided [0.965 to 1.289]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right hand IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5661, MMRM; GLS mean ratio = 1.059, 90% CI 2-sided [0.897 to 1.25]

18. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of ITI as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the duration and variability of ITI for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
seconds
  Left hand ITI variability | 0.036 (0.061) | 0.015 (0.017)
  Right hand ITI variability | 0.053 (0.082) | 0.017 (0.018)
  Left hand ITI duration | 0.064 (0.070) | 0.006 (0.029)
  Right hand ITI duration | 0.094 (0.097) | 0.022 (0.014)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0874, MMRM; GLS mean ratio = 1.571, 90% CI 2-sided [1.018 to 2.424]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.6431, MMRM; GLS mean ratio = 1.18, 90% CI 2-sided [0.644 to 2.162]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left hand ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0389, MMRM; GLS mean ratio = 1.193, 90% CI 2-sided [1.038 to 1.371]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right hand ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1641, MMRM; GLS mean ratio = 1.138, 90% CI 2-sided [0.976 to 1.327]

19. Secondary Outcome: Change From Baseline to Day 28 in the Mean Variability of Peak TF as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The mean changes from Baseline to Day 28 in the variability of TF for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
percentage of variation
  Left hand TF variability | 3.50 (7.44) | 9.98 (2.22)
  Right hand TF variability | 2.5 (10.87) | 3.61 (2.42)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand TF variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5668, MMRM; GLS mean ratio = 0.93, 90% CI 2-sided [0.755 to 1.147]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand TF variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.8686, MMRM; GLS mean ratio = 0.978, 90% CI 2-sided [0.778 to 1.229]

20. Secondary Outcome: Change From Baseline to Day 28 in the Mean Tapping Frequency as Assessed by Dysdiadochomotography
Description: Dysdiadochomotography was used to assess the regularity of hand taps performed when alternating between the palm and dorsal surface of the hand performing a repetitive pronation/supination movement. The force and duration of the hand taps were recorded, with their hand positioned on a force transducer, and recordings were started after practice runs. The patient was then instructed to hand tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each hand. The tapping frequency was calculated as the number of taps between the onsets of the first and the last tap divided by the time in between. The mean changes from Baseline to Day 28 in the tapping frequency for the left and right hands are presented as raw data. GLS mean ratios are in original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 11 | 3
Hertz
  Left hand freq | -0.185 (0.402) | -0.073 (0.088)
  Right hand freq | -0.236 (0.349) | -0.121 (0.189)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left hand freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1244, MMRM; GLS mean ratio = 0.879, 90% CI 2-sided [0.765 to 1.009]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right hand freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3535, MMRM; GLS mean ratio = 0.919, 90% CI 2-sided [0.789 to 1.069]

21. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of IOI as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The mean changes from Baseline to Day 28 in the duration and variability of IOI for the left and right feet are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
seconds
  Left foot IOI variability: number analyzed (Participants) | 9 | 3
  Left foot IOI variability | 0.146 (0.353) | -0.1 (0.122)
  Right foot IOI variability | 0.120 (0.177) | 0.090 (0.15)
  Left foot IOI duration: number analyzed (Participants) | 9 | 3
  Left foot IOI duration | 0.109 (0.354) | -0.123 (0.199)
  Right foot IOI duration | 0.267 (0.461) | 0.075 (0.164)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.015, MMRM; GLS mean ratio = 2.163, 90% CI 2-sided [1.295 to 3.614]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot IOI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.5136, MMRM; GLS mean ratio = 1.274, 90% CI 2-sided [0.688 to 2.361]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left foot IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0218, MMRM; GLS mean ratio = 1.560, 90% CI 2-sided [1.139 to 2.137]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right foot IOI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3720, MMRM; GLS mean ratio = 1.251, 90% CI 2-sided [0.825 to 1.899]

22. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of TD as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The mean changes from Baseline to Day 28 in the duration and variability of TD for the left and right feet are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
seconds
  Left foot TD variability: number analyzed (Participants) | 9 | 3
  Left foot TD variability | 0.225 (0.332) | -0.056 (0.058)
  Right foot TD variability | 0.306 (0.566) | 0.105 (0.140)
  Left foot TD duration: number analyzed (Participants) | 9 | 3
  Left foot TD duration | 0.179 (0.28) | -0.040 (0.106)
  Right foot TD duration | 0.358 (0.609) | 0.083 (0.133)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot TD variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.915, MMRM; GLS mean ratio = 1.911, 90% CI 2-sided [1.017 to 3.592]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot TD variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.2745, MMRM; GLS mean ratio = 1.687, 90% CI 2-sided [0.762 to 3.737]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left foot TD duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1148, MMRM; GLS mean ratio = 1.598, 90% CI 2-sided [0.980 to 2.608]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right foot TD duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3080, MMRM; GLS mean ratio = 1.454, 90% CI 2-sided [0.789 to 2.679]

23. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of IPI as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The mean changes from Baseline to Day 28 in the duration and variability of IPI for the left and right feet are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
seconds
  Left foot IPI variability: number analyzed (Participants) | 9 | 3
  Left foot IPI variability | 0.115 (0.248) | -0.108 (0.131)
  Right foot IPI variability | 0.117 (0.150) | 0.098 (0.164)
  Left foot IPI duration: number analyzed (Participants) | 9 | 3
  Left foot IPI duration | 0.117 (0.383) | -0.123 (0.206)
  Right foot IPI duration | 0.295 (0.469) | 0.073 (0.158)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0079, MMRM; GLS mean ratio = 2.272, 90% CI 2-sided [1.381 to 3.737]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot IPI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0204, MMRM; GLS mean ratio = 1.210, 90% CI 2-sided [0.686 to 2.133]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left foot IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0204, MMRM; GLS mean ratio = 1.564, 90% CI 2-sided [1.144 to 2.138]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right foot IPI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3144, MMRM; GLS mean ratio = 1.269, 90% CI 2-sided [0.856 to 1.884]

24. Secondary Outcome: Change From Baseline to Day 28 in the Mean Duration and Variability of ITI as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The mean changes from Baseline to Day 28 in the duration and variability of ITI for the left and right feet are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day-1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
seconds
  Left foot ITI variability: number analyzed (Participants) | 9 | 3
  Left foot ITI variability | 0.003 (0.203) | -0.047 (0.108)
  Right foot ITI variability | 0.023 (0.118) | -0.016 (0.089)
  Left foot ITI duration: number analyzed (Participants) | 9 | 3
  Left foot ITI duration | -0.049 (0.232) | -0.076 (0.092)
  Right foot ITI duration | -0.016 (0.121) | -0.012 (0.056)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0324, MMRM; GLS mean ratio = 1.914, 90% CI 2-sided [1.167 to 3.141]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot ITI variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.246, MMRM; GLS mean ratio = 1.462, 90% CI 2-sided [0.85 to 2.515]
Statistical Analysis 3: Comparison: BN82451B vs Placebo; Left foot ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1057, MMRM; GLS mean ratio = 1.387, 90% CI 2-sided [0.994 to 1.935]
Statistical Analysis 4: Comparison: BN82451B vs Placebo; Right foot ITI duration statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.7342, MMRM; GLS mean ratio = 1.074, 90% CI 2-sided [0.758 to 1.523]

25. Secondary Outcome: Change From Baseline to Day 28 in the Mean Variability of Peak TF as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The mean changes from Baseline to Day 28 in the variability of TF for the left and right feet are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
percentage of variation
  Left foot TF variability: number analyzed (Participants) | 9 | 3
  Left foot TF variability | 11.63 (16.38) | -20.19 (34.30)
  Right foot TF variability | -2.52 (22.35) | -18.31 (6.52)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot TF variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.1027, MMRM; GLS mean ratio = 1.392, 90% CI 2-sided [0.997 to 1.943]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot TF variability statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.4494, MMRM; GLS mean ratio = 1.158, 90% CI 2-sided [0.840 to 1.595]

26. Secondary Outcome: Change From Baseline to Day 28 in the Mean Tapping Frequency as Assessed by Pedomotography
Description: Pedomotography was used to assess the tap duration and variability in a foot speeded tapping task. The patient placed their foot on the foot device such that the ball of the foot was positioned above a force transducer, and recordings were started after practice runs. The patient was then instructed to foot tap as fast as possible between 2 auditory cues. The beginning of a tap was defined as a rise of the force by 0.05 N above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. 5 trials of 10 seconds duration were performed with each foot. The tapping frequency was calculated as the number of taps between the onsets of the first and the last tap divided by the time in between. The mean changes from Baseline to Day 28 in the tapping frequency for the left and right hands are presented as raw data. The statistical analyses present GLS mean ratios in the original units.
Time Frame: Baseline (Day -1) to Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | BN82451B | Placebo
Number analyzed (Participants) | 10 | 3
Hertz
  Left foot freq: number analyzed (Participants) | 9 | 3
  Left foot freq | -0.259 (0.513) | 0.556 (0.678)
  Right foot freq | -0.383 (0.481) | -0.18 (0.550)
Statistical Analysis 1: Comparison: BN82451B vs Placebo; Left foot freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.0350, MMRM; GLS mean ratio = 0.699, 90% CI 2-sided [0.530 to 0.922]
Statistical Analysis 2: Comparison: BN82451B vs Placebo; Right foot freq statistical analysis is presented (BN82451B versus Placebo). The MMRM analysis was performed on log-transformed data using the REML model including fixed categorical effects of treatment/cohort group, visit and treatment/cohort by visit interaction as well as the continuous fixed covariate of baseline value. Cohort was fitted as random effect; Test type: Superiority or Other; p = 0.3556, MMRM; GLS mean ratio = 0.853, 90% CI 2-sided [0.640 to 1.136]

ADVERSE EVENTS:
Time Frame: From Day 1 to the end of study visit (a period of up to 7 weeks, consisting of up to 28 days of treatment and up to 3 weeks follow up).
Description: AE data is reported as TEAEs.
Arm/Group | BN82451B | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/3
Other Adverse Events (participants affected / at risk) | 11/14 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BN82451B (N=14) | Placebo (N=3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Face oedema (General disorders) | 2 (3) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to subject recruitment problems before the completion of cohort 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not proceed to publication or communication in connection with the subject matter of this Agreement or Results, without the prior written consent of Ipsen.